CLINICAL TRIAL: NCT03205488
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase IIa, Parallel Group, Two Cohort Study to Define the Safety, Tolerability, Clinical and Exploratory Biological Activity of the Chronic Administration of Nilotinib in Participants With Parkinson's Disease
Brief Title: Nilotinib in Parkinson's Disease
Acronym: NILO-PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Rochester (Other); University of Iowa (Other); Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Tanya Simuni, Director, Parkinson's disease and Movement Disorders Center Northwestern University Feinberg School of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NILO-PD
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Results first posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Parkinson Disease
Keywords: Northwestern; Nilotinib; USA; NILO-PD; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Active Comparator): Moderate to Advanced PD Population Randomized 1:1:1
  Interventions: Drug: Cohort 1:Nilotinib Oral Capsules (150mg or 300mg); Drug: Placebo
- Cohort 2 (Active Comparator): Early/de novo Randomized 2:1
  Interventions: Drug: Cohort 2: Nilotinib Oral Capsules (dose to be determined from Cohort 1); Drug: Placebo

INTERVENTIONS:
Drug: Cohort 1:Nilotinib Oral Capsules (150mg or 300mg) — 2 capsules taken once daily
  Arms: Cohort 1
Drug: Cohort 2: Nilotinib Oral Capsules (dose to be determined from Cohort 1) — 2 capsules taken once daily
  Arms: Cohort 2
Drug: Placebo — 2 capsules taken once daily

SUMMARY:
This study will assess the safety and tolerability of daily oral administration of nilotinib (150-300mg once daily) in Parkinson's Disease.

DETAILED DESCRIPTION:
The purpose of this study is to determine if nilotinib is safe, if it can be tolerated by patients with Parkinson's disease (PD) and to learn if nilotinib has the possibility of effectively treating PD symptoms. Nilotinib has been approved by the Food and Drug Administration (FDA) to treat certain types of cancer (leukemia) but is considered investigational in this study because it has not been approved for treating PD. Twenty-five sites will enroll participants into 2 cohorts,approximately 75 in Cohort 1 and 60 in Cohort 2. Participants with moderate to advanced PD symptoms will be enrolled in Cohort 1, randomly assigned to take nilotinib (150 mg or 300mg) or placebo, and will complete 13 in-person study visits over 8.5 months.

The results from Cohort 1 will determine if either dose of nilotinib (150mg or 300 mg) is safe and tolerable enough to move forward and evaluate in Cohort 2. If either dose is found to be safe and tolerable, participants with early PD will be enrolled into Cohort 2.

Participants in Cohort 2 will be randomly assigned to either nilotinib (dose to be determined from Cohort 1 results) or placebo and will complete 17 in-person visits over 14.5 months. For both cohorts, the study visits will include clinical assessment of motor, neuropsychiatric and cognitive testing as well as collection of blood and cerebral spinal fluid, collected by lumbar puncture.

This study will also evaluate if nilotinib can help improve motor symptoms associated with PD. All participants in Cohort 1 and participants in Cohort 2 who have started PD medications will have an assessment of the motor exam (Part III) in a practically defined OFF state (12 hours post dose) and ON state (at least one-hour post dose).

ELIGIBILITY:
Inclusion Criteria; Cohort 1 and 2:

1. Idiopathic PD based on the UK Brain Bank diagnostic criteria.
2. Any race and either gender, age 40-79
3. Able to read and understand English with the capacity to provide voluntary informed consent by signing the informed consent form (ICF)
4. Willing to comply with all study procedures including multiple lumbar punctures (LP)
5. Must be on a stable regimen of central nervous system acting medications (if applicable) for at least 30 days prior to the baseline visit (e.g., benzodiazepines, antidepressants, hypnotics)

Inclusion criteria specific for Cohort 1:

6a. Diagnosis of PD duration > 5 year 7a. Hoehn & Yahr scale (H&Y) stage > 2 and < 4 in the ON state 8a. Must be on a stable regimen of PD medications, that includes levodopa, for at least 30 days prior to the screening visit

a. Treatment with monoamine oxidase B (MAO-B) inhibitors will be allowed provided the dose has been stable for 60 days prior to baseline

Inclusion criteria specific for Cohort 2:

6b. Diagnosis of PD duration < 3 years 7b. H&Y stage ≤ 2 8b. Participants who are currently NOT receiving symptomatic therapy (ST) (levodopa,dopamine agonists and monoamine oxidase B (MAO-B) inhibitors) and NOT projected to require ST for at least 3 months from enrollment.

a. Treatment with amantadine or an anticholinergic agent will be allowed provided the dose has been stable for 30 days prior to screening and will remain stable for the duration of the study

Exclusion Criteria; Cohorts 1 and 2:

1. Diagnosis of atypical parkinsonism
2. History of bipolar disorder or major depression, or presence of active depression defined as a Beck Depression Inventory II (BDI-II) score >17
3. History of a suicide attempt within the last 5 years or active suicidal ideations
4. History of schizophrenia or schizophrenia spectrum disorders
5. History of uncontrolled hypokalemia or hypomagnesaemia, or laboratory evidence of such on screening
6. History of cardiac arrhythmia, long QT syndrome, or a corrected QT interval (QTcF) ≥450ms at screening visit 1
7. Treated within 30 days prior to randomization, or planned use during the trial with any of the following classes of Concomitant drugs:

   1. Class IA or III antiarrhythmic drugs
   2. QT prolonging drugs
   3. Strong CYP3A4 inhibitors or inducers
   4. Anticoagulants
   5. Proton pump inhibitors
8. A clinical history, or the active presence of a cardiovascular condition including:

   1. Myocardial infarction, known cardiac ischemia, or angina
   2. Cerebrovascular event (e.g. embolic stroke)
   3. Congestive heart failure, symptomatic first degree atrioventricular (AV) block or PR interval > 220msec and all second and third degree AV block, second- or third-degree atrioventricular block, sick sinus syndrome, or other serious cardiac rhythm disturbances
   4. History of Torsade de Pointes
   5. Other cardiovascular history that, in the opinion of the Site Investigator, will preclude study participation
9. History of hepatic disease, including abnormal liver function defined as Total Bilirubin > 1.5 times upper limit, Aspartate Aminotransferase (AST) and/or Alanine Aminotransferase (ALT) > 2 times the upper limit of the normal, or coagulopathy with INR > 1.4
10. History of epilepsy or a seizure within the last 6 months
11. Active malignancy, or history of a neoplasm in the prior 5 years (excluding basal/squamous cell carcinoma)
12. Prior history of pancreatitis or total gastrectomy or evidence of abnormal pancreatic function defined as elevated amylase and/or lipase > 2 times upper limit of normal
13. Diagnosis of human immunodeficiency virus (HIV), clinically significant chronic hepatitis such as hepatitis B (HBV) or hepatitis C (HCV), or clinical history or signs of an active infection
14. History of drug or alcohol abuse ≤ 5 years
15. Active medical or psychiatric condition that in the opinion of the Site Investigator should preclude study participation
16. Previous surgical management for PD
17. Participants participating in any drug or device clinical investigation concurrently or within 30 days prior to screening for this study
18. Severe lactose and galactose intolerance
19. Participants with evidence of other significant laboratory abnormalities which in the opinion of the site investigator or clinical monitor should preclude study participation
20. Known hypersensitivity or contraindication to study drugs (nilotinib or matching placebo) or their components.
21. Female participants of child-bearing potential. Female participants must be post-menopausal, post-hysterectomy, or have a documented infertility based on a known medical or surgical condition
22. Participants with a history of bone marrow suppression or evidence of persistent myelosuppression defined as absolute neutrophil count <1.8 X 109/L, significant anemia, or thrombocytopenia defined as platelet count < 100 X 109/L

Exclusion criteria specific for Cohort 1:

22a. Diagnosis of dementia based on the clinician's assessment, or a Montreal Cognitive Assessment (MoCA) score < 21 at baseline

Exclusion criteria specific for Cohort 2:

22b.MoCA score < 26 at baseline 23b. Treated within 60 days prior to randomization or expected to require treatment within 3 months from randomization with any ST (including levodopa and dopamine agonists )

a. Treatment with amantadine or an anticholinergic agent will be allowed provided the dose has been stable for 30 days prior to screening and will remain stable for the duration of the study

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Simuni, MD, Principal Investigator — Northwestern University
Locations (24):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Sun City, Arizona
  - University of California Davis, Sacramento, California
  - University of Colorado at Denver, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - John Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Cleveland Clinic - Las Vegas, Las Vegas, Nevada
  - Albany Medical College, Albany, New York
  - Beth Israel Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inland Northwest Research, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joshi D, Kulkarni M, Parekh P, Shah S, Greig NH, Acharya S. Targeting protein kinases in Parkinson's disease: the emerging role of phytoconstituents. Nutr Neurosci. 2025 Dec;28(12):1532-1563. doi: 10.1080/1028415X.2025.2531356. Epub 2025 Jul 18. PMID 40680102
- [Derived] Simuni T, Fiske B, Merchant K, Coffey CS, Klingner E, Caspell-Garcia C, Lafontant DE, Matthews H, Wyse RK, Brundin P, Simon DK, Schwarzschild M, Weiner D, Adams J, Venuto C, Dawson TM, Baker L, Kostrzebski M, Ward T, Rafaloff G; Parkinson Study Group NILO-PD Investigators and Collaborators. Efficacy of Nilotinib in Patients With Moderately Advanced Parkinson Disease: A Randomized Clinical Trial. JAMA Neurol. 2021 Mar 1;78(3):312-320. doi: 10.1001/jamaneurol.2020.4725. PMID 33315105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From November 2017 to December 2018, 125 patients were assessed for eligibility. Of those screened, 76 participants were enrolled in the trial.
Pre-assignment Details: Of the patients assessed for eligibility, 49 (39%) were excluded. 42 patients did not meet inclusion criteria and 7 declined study participation.
Groups:
- Placebo: Placebo enclosed in capsules to maintain the blind was administered orally once per day over the course of 6 months.
- Nilotinib 150: Patients were administered 1 capsule of 150 mg Nilotinib and 1 capsule of matching placebo each day over the course of 6 months.
- Nilotinib 300: Patients were administered 2 capsules of 150 mg Nilotinib each day over the course of 6 months.
Period: Overall Study
Arm/Group | Placebo | Nilotinib 150 | Nilotinib 300
Started | 25 | 25 | 26
Completed | 24 | 23 | 21
Not Completed | 1 | 2 | 5
Not completed — Adverse Event | 1 | 2 | 4
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nilotinib 150 | Nilotinib 300 | Total
Number analyzed (Participants) | 25 | 25 | 26 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 16 | 9 | 38
  >=65 years | 12 | 9 | 17 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (6.8) | 61.2 (7.4) | 66.9 (7.3) | 64.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 5 | 24
  Male | 16 | 15 | 21 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 24 | 25 | 25 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 24 | 23 | 25 | 72
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 26 | 76
Parkinson's Disease History [Mean (Standard Deviation); unit: years]
  Parkinson's Disease Duration | 9.4 (4.9) | 8.5 (3.2) | 11.7 (5.2) | 9.9 (4.7)
  Age at Diagnosis | 56.2 (6.8) | 52.7 (7.6) | 55.2 (9.3) | 54.7 (8.0)
MDS-UPDRS Total Score [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Baseline total Unified Parkinson Disease Rating Scale (UPDRS) score ranges from 0 to 295. The higher the value the more disability from PD the participant has.
  units on a scale
    MDS-UPDRS Total OFF Score | 63.8 (21.3) | 65.0 (16.0) | 70.2 (20.2) | 66.4 (19.3)
    MDS-UPDRS Total ON Score | 46.2 (17.8) | 46.9 (15.1) | 51.9 (15.7) | 48.4 (16.2)
Parkinson's Disease Classifications [Count of Participants; unit: Participants] — Measure Description: Hoehn and Yahr staging of severity of Parkinson's disease. Baseline H/Y stage ranges from >2 to <4. Larger value stands for more disability from PD. H&Y 2 = Bilateral involvement without impairment of balance. H&Y 3 = Mild to moderate involvement; some postural instability but physically independent; needs assistance to recover from pull test. 4 = Severe disability; still able to walk or stand unassisted.
  Participants
    Hoehn and Yahr Stage 0-2 | 4 | 5 | 1 | 10
    Hoehn and Yahr Stage 3 | 21 | 20 | 25 | 66
    Class of Symptomatic Therapy, MAOB Inhibitors | 11 | 8 | 12 | 31
Levodopa Equivalent Daily Dose [Mean (Standard Deviation); unit: mg] | 1066.5 (519.7) | 971.8 (251.4) | 1012.5 (390.5) | 1016.9 (398.7)
Education Adjusted MoCA Score [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Montreal Cognitive Assessment (MoCA) is one-page 30-point test to detect cognitive impairment. Baseline MoCA score ranges from 23 to 30. Higher scores indicate better cognition.
  units on a scale | 26.9 (2.4) | 27.4 (1.9) | 27.0 (2.4) | 27.1 (2.2)
DRS-2 [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Mattis Dementia Rating Scale 2 (DRS-2) is a test to screen for dementia in Parkinson's disease. Five subscales provide additional information on specific abilities: Attention, Initiation/Perseveration, Construction, Conceptualization, and Memory. DRS-2 score range is 0-144. Higher scores indicate better cognition.
  units on a scale | 138.1 (5.7) | 137.8 (7.8) | 137.7 (6.3) | 137.9 (6.6)
BDI-II [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Baseline Beck Depression Inventory (BDI) score ranges from 0 to 23. Higher scores indicate greater symptom severity.
  units on a scale | 6.6 (4.9) | 7.3 (5.4) | 6.6 (4.3) | 6.8 (4.8)
PDSS [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Parkinson Disease Sleep Scale self-rate and quantify the level of sleep disruption being experienced in order to target treatment appropriately. Scores range from 0 to 150. Higher scores indicate greater symptom severity.
  units on a scale | 106.6 (21.8) | 115.3 (11.6) | 103.2 (18.6) | 108.3 (18.3)
Modified S/E ADL [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Schwab and England Activities of Daily Living scale. Baseline SE/ADL ranges from 40 to 100. Smaller value stands for more disability from PD.
  units on a scale
    Modified S/E ADL OFF | 73.2 (16.5) | 77.3 (17.8) | 77.0 (14.9) | 75.8 (16.8)
    Modified S/E ADL ON | 86.8 (8.7) | 92.2 (5.8) | 87.0 (17.9) | 88.6 (12.2)
PDQ-39 [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Parkinson's Disease Questionnaire-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the past month. Baseline PDQ 39 score ranges from 0 to 52. Lower score shows better quality of life.
  units on a scale | 19.0 (12.7) | 19.0 (9.4) | 18.4 (10.3) | 18.8 (10.8)
EQ-5D [Mean (Standard Deviation); unit: units on a scale] — Measure Description: EQ-5D summary index is derived by applying a formula that essentially attaches values (weights) to each of the levels in the 5 dimensions. The total index range is from 0-1. The Health Score range is 0-100 point scale where the participant marks his or her health related quality that day. Higher scores show better quality of life.
  units on a scale
    EQ-5D Summary Index | 0.79 (0.14) | 0.83 (0.13) | 0.78 (0.15) | 0.80 (0.14)
    EQ-5D Health Score | 70.6 (25.1) | 71.5 (23.3) | 76.0 (15.9) | 72.8 (21.5)

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of Nilotinib Over Placebo
Description: The count of study participants who completed the 6-month study treatment period while active on their original assigned dose
Time Frame: 6 months
Population: Intent-to-treat population, all randomized subjects per arm. The Count of participants below are the number of participants that met the criteria for analysis of tolerability.
Measure: Count of Participants; unit: Participants
Groups:
- Nilotinib 150 mg: Patients were administered 1 capsule of 150 mg Nilotinib and 1 capsule of matching placebo each day over the course of 6 months.
- Nilotinib 300 mg: Patients were administered 2 capsules of 150 mg Nilotinib each day over the course of 6 months.
Arm/Group | Placebo | Nilotinib 150 mg | Nilotinib 300 mg
Number analyzed (Participants) | 25 | 25 | 26
Participants | 21 | 19 | 20
Statistical Analysis 1: Comparison: Placebo vs Nilotinib 150 mg; Test type: Superiority; p = 0.3626, Fisher Exact; One-sided Fisher's Exact tested the proportion of participants who met tolerability between the Nilotinib 150 group to the Placebo group
Statistical Analysis 2: Comparison: Placebo vs Nilotinib 300 mg; Test type: Superiority; p = 0.3895, Fisher Exact; One-sided Fisher's Exact tested the proportion of participants who met tolerability between the Nilotinib 300 group to the Placebo group

2. Primary Outcome: Safety of Nilotinib
Description: The count of study participants who experienced any treatment-related SAE in each treatment group
Time Frame: We assessed adverse events that were collected from the first dose of study drug until 60 days after the participant's last dose.
Population: Intent-to-treat population, all randomized subjects. The counts refer to the number of participants that experienced an SAE in each treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nilotinib 150 | Nilotinib 300
Number analyzed (Participants) | 25 | 25 | 26
Participants | 2 | 1 | 1
Statistical Analysis 1: Comparison: Placebo vs Nilotinib 150; Test type: Equivalence — H0 : p1 = p2, where p represents the proportion of SAEs for each group. HA : p1 ≠ p2; p = 1.00, Fisher Exact; Fisher's Exact test compared a proportion of participants who experienced any serious adverse event in the Nilotinib 150 group and the Placebo group
Statistical Analysis 2: Comparison: Placebo vs Nilotinib 150; Test type: Equivalence — H0 : λ1 = λ2, where λ represents the rate of SAEs for each group. HA : λ1 ≠ λ2; p = 0.5689, Regression, Poisson; Rates of serious adverse event between the Nilotinib 150 group and the placebo were also compared using a Poisson regression model; Risk Ratio (RR) = 0.4977, 95% CI 2-sided [0.0451 to 5.489]
Statistical Analysis 3: Comparison: Placebo vs Nilotinib 300; Test type: Equivalence — H0 : p1 = p3, where p represents the proportion of SAEs for each group. HA : p1 ≠ p3; p = 0.61, Fisher Exact; Fisher's Exact test compared a proportion of participants who experienced any serious adverse event in the Nilotinib 300 group and the Placebo group
Statistical Analysis 4: Comparison: Placebo vs Nilotinib 300; Test type: Equivalence — H0 : λ1 = λ3, where λ represents the rate of SAEs for each group. HA : λ1 ≠ λ3; p = 0.5940, Regression, Poisson; Rates of serious adverse event between the Nilotinib 300 group and the placebo were also compared using a Poisson regression model; Risk Ratio (RR) = 0.5206, 95% CI 2-sided [0.0472 to 5.7409]

3. Secondary Outcome: Change in MDS-UPDRS Part III
Description: The Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III is a motor examination in both practically defined medications OFF state (12 hrs post dose) and ON state (based on the participant/site investigator defined best ON and/or approximately 1 hour post dose). Measure Description: The part III subscale score ranges from 0-165. The Larger the value stands for more disability from PD.
Time Frame: The MDS-UPDRS Part III ON state was collected at baseline, day 14, day 30, month 3, month 6, 30 and 60 days post treatment. The OFF state was collected at baseline, month 3, month 6, 30 and 60 days post treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo enclosed in capsules to maintain the blind was administered orally twice per day over the course of 6 months.
Arm/Group | Placebo | Nilotinib 150 | Nilotinib 300
Number analyzed (Participants) | 25 | 25 | 26
units on a scale
  Baseline MDS-UPDRS Part III (ON) | 22.80 (8.85) | 24.76 (11.62) | 25.15 (8.17)
  Day 14 MDS-UPDRS Part III (ON) | 23.13 (11.29) | 27.58 (13.53) | 29.33 (9.77)
  Day 30 MDS-UPDRS Part III (ON) | 22.36 (10.00) | 26.84 (13.08) | 29.73 (10.83)
  Month 3 MDS-UPDRS Part III (ON) | 19.83 (9.23) | 24.88 (13.70) | 25.76 (8.71)
  Month 6 MDS-UPDRS Part III (ON) | 19.63 (9.86) | 24.43 (11.50) | 25.61 (8.93)
  30 Day Post MDS-UPDRS Part III (ON) | 20.52 (8.82) | 25.13 (12.26) | 26.79 (9.10)
  60 Day Post MDS-UPDRS Part III (ON) | 20.88 (10.88) | 23.91 (12.93) | 26.42 (10.58)
  Baseline MDS-UPDRS Part III (OFF) | 40.36 (13.51) | 42.84 (12.53) | 43.50 (14.01)
  Month 3 MDS-UPDRS Part III (OFF) | 37.92 (14.46) | 39.92 (12.41) | 41.04 (13.38)
  Month 6 MDS-UPDRS Part III (OFF) | 36.21 (14.91) | 41.91 (13.40) | 43.96 (11.62)
  30 Day Post MDS-UPDRS Part III (OFF) | 38.92 (14.15) | 41.48 (12.19) | 45.26 (14.13)
  60 Day Post MDS-UPDRS Part III (OFF) | 37.36 (14.20) | 40.27 (11.33) | 43.00 (13.63)
Statistical Analysis 1: Comparison: Placebo vs Nilotinib 150; The key secondary objective is to conduct a futility analysis within each treatment group which examines the observed change in the MDS-UPDRS Part III ON within the two dose groups compared to previously reported changes from the Pagan et al (2016) study (NCT02281474); Test type: Non-Inferiority — The hypotheses of interest (H0: δ ≤ -9.8 (7 x 1.4) vs. HA: δ > -9.8) where δ represents the change from baseline to 6 months using the MDS-UPDRS Part III ON in the Nilotinib 150 mg treatment group. The hypotheses of interest were evaluated based on an assessment of parameter estimates from a non-linear mixed effects model, adjusted for a participant's Levodopa Equivalent Daily Dose (LEDD) at each time point; p = 0.0001, Mixed Models Analysis; Slope = 1.05, 90% CI 1-sided [lower limit -0.78]
Statistical Analysis 2: Comparison: Placebo vs Nilotinib 300; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority — The hypotheses of interest (H0: δ ≤ -9.8 (7 x 1.4) vs. HA: δ > -9.8) where δ represents the change from baseline to 6 months using the MDS-UPDRS Part III ON in the Nilotinib 300 mg treatment group. The hypotheses of interest were evaluated based on an assessment of parameter estimates from a non-linear mixed effects model, adjusted for a participant's Levodopa Equivalent Daily Dose (LEDD) at each time point; p = 0.0001, Mixed Models Analysis; Slope = 0.93, 90% CI 1-sided [lower limit -0.89]
Statistical Analysis 3: Comparison: Placebo vs Nilotinib 150 vs Nilotinib 300; Additional secondary objective #1 is to establish the degree of symptomatic effect of Nilotinib as measured by the change in the MDS_UPDRS Part III ON score between baseline and 1 month; Test type: Equivalence — H0 : β1 = β 2 = β 3, where β represents the slope for each group. HA : at least one β i ≠ β j. Using the same LMM as in the key secondary analysis, a two degree of freedom test was used to test for any differences in the slopes from baseline to 1 month for the three treatment groups; p = 0.031, Mixed Models Analysis; In order to assess which group may be driving these findings, pairwise comparisons were also utilized (Nilotinib 150 vs PBO at 1 Month, Nilotinib 300 vs PBO at 1 month, Nilotinib 300 vs Nilotinib 150 at 1 month)
Statistical Analysis 4: Comparison: Placebo vs Nilotinib 150 vs Nilotinib 300; Additional secondary objective #2 is to establish the degree of symptomatic effect of Nilotinib as measured by the change in the MDS_UPDRS Part III ON score between the final visit on study drug and 30 days off study drug; Test type: Equivalence — H0 : β1 = β 2 = β 3, where β represents the slope for each group. HA : at least one β i ≠ β j. For this analysis, a separate LMM was constructed, modeling the change from final visit on study drug to the 30 and 60 day follow up visits, while adjusting for the MDS-UPDRS Part III ON scores at the final visit on study drug as well as the Levodopa Equivalent Daily Dose (LEDD) at each visit; p = 0.47, Mixed Models Analysis
Statistical Analysis 5: Comparison: Placebo vs Nilotinib 150 vs Nilotinib 300; Additional secondary objective #3 is to assess the impact of Nilotinib on the progression of PD disability as measured by the change in the MDS_UPDRS Part III ON score between baseline and 6 months; Test type: Equivalence — H0 : β1 = β 2 = β 3, where β represents the slope for each group. HA : at least one β i ≠ β j. Using the same LMM as in the key secondary analysis, a two degree of freedom test was used to test for any differences in the slopes from baseline to 6 months for the three treatment groups; p = 0.077, Mixed Models Analysis; Pairwise comparisons were also examined for trends (Active 150 vs PBO at 6 Months, Active 300 vs PBO at 6 months)
Statistical Analysis 6: Comparison: Placebo vs Nilotinib 150 vs Nilotinib 300; Additional secondary objective #3 is to assess the impact of Nilotinib on the progression of PD disability as measured by the change in the MDS_UPDRS Part III OFF score between baseline and 6 months; Test type: Equivalence — H0 : β1 = β 2 = β 3, where β represents the slope for each group. HA : at least one β i ≠ β j. Using a similar LMM as in the key secondary analysis, except simplified to only include baseline, month 3 and month 6, a two degree of freedom test was used to test for any differences in the slopes from baseline to 6 months for the three treatment groups; p = 0.17, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected following the first dose of study drug until 30 days after the participant's last dose of study drug.
Groups:
- Nilotinib 150: Patients were administered 1 capsule of 150 mg Nilotinib and 1 capsule of matching placebo once per day over the course of 6 months.
- Nilotinib 300: Patients were administered 2 capsules of 150 mg Nilotinib once per day over the course of 6 months.
Arm/Group | Placebo | Nilotinib 150 | Nilotinib 300
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 2/25 | 1/25 | 1/26
Other Adverse Events (participants affected / at risk) | 22/25 | 23/25 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Nilotinib 150 (N=25) | Nilotinib 300 (N=26)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Nilotinib 150 (N=25) | Nilotinib 300 (N=26)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (5)
Fatigue (General disorders) | 4 (5) | 4 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 2 (2) | 2 (3)
Urinary tract infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Amylase Increased (Investigations) | 2 (2) | 4 (4) | 4 (6)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
CSF protein increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 4 (5) | 7 (11) | 6 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)
Tremor (Nervous system disorders) | 1 (2) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (11) | 4 (4) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/88/NCT03205488/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT03205488/SAP_001.pdf